CLINICAL TRIAL: NCT05631912
Title: Autologous TRAC Locus-inserted CD19-targeting Synthetic T-cell Receptor Antigen Receptor T (STAR-T) Cells for Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: TRAC Locus-inserted CD19-targeting STAR-T Cell Therapy in r/r B-NHL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-073
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Non-hodgkin Lymphoma,B Cell
MeSH Terms: interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous TRAC locus-inserted CD19-targeting STAR-T cells (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide (FC regimen) will be administered followed by investigational treatment, autologous targeting CD19 synthetic T-cell receptor antigen receptor T cells.
  Post leukapheresis, administration of short half-life chemo-agents, Bruton tyrosine kinase inhibitor (BTKi) and/or dexamethasone should be considered to bridge the following FC regimen in patients with bulky tumor burden, rapidly aggressive progression, and/or indications of imperious symptom control.
  Interventions: Biological: Autologous CD19-STAR-T cell; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Autologous CD19-STAR-T cell — Phase 1 dose escalation (3+3) : dose 1 (1×10^6 cells/kg) ,dose 2 (3×10^6 cells/kg) ,dose 3 (1×10^7 cells/kg); Phase 2 : Appropriate dose
  Other Names: Autologous CD19-targeting synthetic T-cell receptor antigen receptor T cells
Drug: Fludarabine — Intravenous fludarabine 25-30 mg/m^2/day on days -5, -4, and -3.
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide 300-500 mg/m^2/day on days -5, -4, and -3.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
The team has developed a chimeric antigen receptor (CAR) based on T cell receptor (TCR) complex, called synthetic TCR and antigen receptor (STAR). Further, the researchers disrupted the endogenous T-cell receptor α constant (TRAC) locus by CRISPR/cas9, and then knocked in the anti-CD19-STAR construct through TRAC endogenous promoter. In this single center, prospective, open-label, single-arm, phase 1/2 study, the safety and efficacy of autologous CD19-targeting STAR-T cell therapy will be evaluated in patients with relapsed or refractory (r/r) B-cell non-Hodgkin's lymphoma (B-NHL) . A total of 19 to 38 patients are planned to be enrolled and receive CD19-STAR-T cell infusion. Phase 1 (9 to 18 cases) is dose escalation part, and phase 2 (10 to 20 cases) is expansion cohort part.

DETAILED DESCRIPTION:
[Introduction]

At present, CAR-T cell therapy targeting CD19 has achieved remarkable efficacy in the treatment of r/r B-NHL. However, at the same time, CAR-T cell treatment has a high incidence of cytokine release syndrome (CRS), immune cell-associated neurotoxicity syndrome (ICANS) and other toxicities. TCR-T is another adoptive T cell therapy, which recognizes the surface and intracellular antigens of target cells presented by major histocompatibility complex (MHC) molecules and engage CD3 signaling machinery, triggering a wide range of TCR-CD3 signaling to kill tumors. TCR-T is characterized by high affinity with target antigen, low toxicity, but difficulty in preparation.

Here, the researchers connected the murine TCR constant regions α and β with the light chain and heavy chain of the murine FMC63 single-chain variable fragment (scFv) respectively to construct a human leukocyte antigen (HLA)-independent antibody TCR chimera, called synthetic T cell receptor and antigen receptor (STAR). Then, researchers introduced an additional interchain disulfide bond by making cysteine mutations within TCRα/β constant regions, and employed hydrophobic substitutions to the TCR-α chain transmembrane domain to improve the receptor's stability on plasma membrane.

Further, the team disrupted the endogenous TRAC locus by CRISPR/cas9, and then knocked in the CD19-STAR construct to this locus, and transcription of CD19-STAR triggered by the TRAC endogenous promoter. TRAC locus knockout can prevent endogenous TCR assembly, and avoid the harm caused by graft-versus host disease (GVHD) as well as random insertion. This specific integration of "two in one" technology can give rise to highly efficient expression of CD19-STAR chimeric molecule on T cell surface, and the subsequent assembly of complete TCR signaling structure.

The molecular structure of STAR in this study: the variable region of TCRα/β chain is replaced with the heavy chain and light chain of FMC63 antibody respectively, the intracellular region of α/β chain is connected with an OX40 costimulatory molecule respectively.

STAR integrates the advantages of TCR and CAR, and is close to the natural TCR-antigen action mode with high affinity, high sensitivity, and low T cell exhaustion. Compared with TCR-T, it is easier to obtain and prepare. The researchers confirmed that the CD19-STAR-T cells, by in vitro and in vivo assays, had lower cytokine release but more efficient anti-tumor activities when compared to canonical CAR-T cells. In this study, we would like to evaluate the safety and efficacy of autologous TRAC locus-inserted CD19-STAR-T cell in r/r patients with r/r B-NHL . The completion of this trial will provide a research foundation for potential universal allogeneic adoptive T cell therapy.

[Study design]

Phase 1 (dose escalation)

In phase 1, 9 to 18 subjects will be enrolled. Subjects will receive 3 doses of CD19-STAR-T cell therapy (1 × 10^6 cells/kg, 3 × 10^6 cells/kg, 1 × 10^7 cells/kg) from low dose to high dose according to the "3 + 3" principle:

1. Three patients were enrolled in the lowest dose group.
2. Subsequent patients were enrolled according to the following rules:

   1. If the incidence of dose limiting toxicity (DLT) was 0/3, 3 patients were enrolled in the next high-dose group.
   2. If the incidence of DLT was 1/3, 3 patients were enrolled at the same dose; If the incidence of DLT was 1/3 + 0/3, 3 patients were enrolled in the next high-dose group. If the incidence of DLT was 1/3 + 1/3, this dose was defined as maximum tolerated dose (MTD); If the incidence of DLT was 1/3 + 2/3 or 1/3 + 3/3, the previous dose was MTD.
   3. If the incidence of DLT was 2/3 or 3/3, the previous dose was MTD.

To ensure the safety of the subjects, the first subject in each dose group was observed for at least 28 days after the cell infusion. If no DLT occurred, the remaining two subjects could be enrolled and treated at the same dose level. The safety data of all subjects in each dose group until day 28 should be reviewed and tolerated before proceeding to the next dose group trial. No dose escalation was allowed for the same subject during the trial. If a subject drop out during the observation period due to non-DLT reasons, new subjects should be enrolled to make up for the number of subjects who drop out.

Phase 2 (expansion cohort)

In phase 2, 10 to 20 subjects will be enrolled and receive CD19-STAR-T cell infusion at dose of RP2D, which will be determined based on the MTD, occurrence of DLT, the obtained efficacy results, pharmacokinetics / pharmacodynamics and other data according to the phase 1.

[Objectives]

The primary objectives of the phase 1 were to evaluate the tolerability, safety, and determine recommended phase 2 dose (RP2D). The primary purpose of the phase 2 study was to evaluate the efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (inclusive).
2. Patients with histologically confirmed CD19-positive B-cell NHL, including the following types defined by the World Health Organization (WHO) 2016:

   * Diffuse large B-cell lymphoma not otherwise specified (DLBCL-NOS), including Activated B-cell type (ABC) / Germinal center B-cell Type (GCB);
   * Primary mediastinal (thymic) large B-cell lymphoma (PMBCL);
   * Transformed follicular lymphoma (TFL);
   * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements (HGBCL);
   * Follicular lymphoma (FL);
   * Mantle cell lymphoma (MCL) [pathologically confirmed, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1];
   * Marginal zone lymphoma (MZL), including nodal or splenic marginal zone B-cell lymphoma and mucosa-associated lymphoid tissue (MALT) lymphoma.
3. Relapse after treatment with ≥2 lines systemic therapy for all the above disease types, or refractory disease for aggressive types (DLBCL-NOS, PMBCL, TFL and HGBCL). Relapse disease is defined as disease progression after last regimen. Refractory disease is defined as no CR to first-line therapy:

   * PD as best response to first-line therapy, or
   * SD as best response after at least 4 cycles of first-line therapy (eg, 4 cycles of R-CHOP), or
   * PR as best response after at least 6 cycles and biopsy-proven residual disease or disease progression ≤ 6 months of therapy, or
   * Refractory post-autologous stem cell transplant (ASCT) i. Disease progression or relapsed less than or equal to 12 months of ASCT (must have biopsy proven recurrence in relapsed individuals) ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy.
4. Individuals must have received adequate prior therapy:

   * For MCL, prior therapy must have included:

     * Anthracycline or bendamustine-containing chemotherapy and
     * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
     * Bruton's tyrosine kinase inhibitor (BTKi)
   * For other types, prior therapy must have included:

     * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
     * Anthracycline containing chemotherapy regimen.
   * For individual with transformed FL must have relapse or refractory disease after transformation to DLBCL.
5. The estimated survival time is over 3 months.
6. The Eastern Cooperative Oncology Group (ECOG) score is 0-2.
7. According to Lugano response criteria 2014, there should be at least one evaluable tumor focus. Evaluable tumor focus was defined as that with the longest diameter of intranodal focus > 1.5cm, the longest diameter of extranodal focus > 1.0cm assessed by computed tomography (CT) or magnetic resonance imaging (MRI).
8. Subjects must be willing to undergo either excised or large-needle lymph node or tissue biopsy, or provide formalin-fixed paraffin-embedded (FFPE) tumor tissue block or freshly cut unstained slides.
9. Functions of important organs meet the following requirements: Echocardiography showed left ventricular ejection fraction ≥50%. Serum creatinine ≤1.5 × upper limit of normal range (ULN) or endogenous creatinine clearance ≥45mL/min (cockcroft-gault formula); Alanine ULN, Total bilirubin ≤1.5× ULN; Pulmonary function: ≤CTCAE grade 1 dyspnea and oxygen saturation of blood (SaO2) ≥91% in indoor air environment.
10. Blood routine (normal values shall not be obtained with growth factors, and hemocytopenia caused by lymphoma invasion of bone marrow is not subject to conditions below): hemoglobin (Hgb) ≥80g/L, neutrophil count (ANC) ≥1×10^6/L, platelet (PLT) ≥75×10^9/L.
11. Pregnancy tests for women of childbearing age shall be negative; Both men and women agreed to use effective contraception during treatment and during the subsequent 1 year.
12. Toxicity from previous antitumor therapy ≤ grade 1 (according to CTCAE version 5.0) or to an acceptable level of inclusion/exclusion criteria (other toxicities such as alopecia and vitiligo considered by the investigator to pose no safety risk to the subject).
13. No obvious hereditary diseases.
14. Able to understand the requirements and matters of the trial, and willing to participate in clinical research as required.
15. Informed consent must be signed.

Exclusion Criteria:

1. During the screening period, there was central nervous system (CNS) invasion or a history of clinically significant central nervous system diseases, such as epilepsy and cerebrovascular diseases.
2. Women who are pregnant or breastfeeding, or who do not agree to use effective contraception during treatment and during the subsequent 1 year.
3. History of allogeneic hematopoietic stem cell transplantation, or organ transplantation.
4. History of other malignancies that have not been in remission.
5. Patients with primary immunodeficiency or autoimmune diseases requiring immunosuppressive therapy.
6. Received radiotherapy within 3 months before enrollment.
7. Received immunotherapy drugs within 4 weeks before enrollment, such as anti-programmed death 1 (PD-1) antibody, anti-programmed death ligand 1 (PD-L1) antibody, CD19/CD3-bispecific antibody, and so on.
8. Patients who received any immunocellular therapy within 6 months before enrollment.
9. Confirmed evidence showing positiveness of anti-CD19 scFv reaction in patient serum.
10. Patients who participated in other clinical trials within 4 weeks prior to enrollment.
11. Uncontrolled infectious diseases or other serious illnesses, including but not limited to infections [e.g., human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B (HBV) or C (HCV) infection], congestive heart failure, unstable angina, arrhythmias, or that pose an unpredictable risk in the opinion of the attending physician.
12. The presence of uncontrollable serous membrane fluid, such as massive pleural effusion or ascites.
13. A history of stroke or intracranial hemorrhage within 3 months prior to enrollment.
14. Major surgery or trauma occurred within 28 days prior to enrollment, or major side effects have not been recovered.
15. History of allergies to any of the ingredients in cell products.
16. Conditions in which a known mental or physical illness interferes with cooperation with the requirements of the study or disrupts the results or interpretation of the results and, in the opinion of the therapeutic investigator, makes the patient unfit for study participation.
17. There is the situation that the researcher's judgment will interfere with the whole study participation; Situations where there is significant risk to the subject; Or interferes with the interpretation of research data.
18. Inability to understand or unwillingness to sign informed consent.
19. Researchers believe that other reasons are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of Adverse Events (AEs) | 12 months
  AE is defined as any adverse medical event from the date of randomization to 12 months after CD19-STAR-T cells infusion. Among them, CRS and ICANS were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
Phase 1: Incidence of Dose-Limiting Toxicities (DLTs) | First infusion date of CD19-STAR-T cells up to 28 days
  DLT was defined as CD19-STAR-T cells-related events with onset within first 28 days following infusion: The development of Grade (G) 3 or higher grade CRS lasting > 2 weeks; Any CD19-STAR-T cells-related AE requiring intubation; All G4 non-hematologic toxicities.
Phase 1: Maximum tolerated dose (MTD) | 12 months
  MTD is defined as the highest dose level of less than or equal to 2 DLT among the 6 subjects finally determined.
Phase 1: Recommended phase 2 dose (RP2D) | 12 months
  The recommended dose for phase 2 was determined through phase 1 study.
Phase 2: Best objective Response Rate | 12 months
  The incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as the best response to treatment assessed by investigators and based on the Lugano 2014 assessment criterion.

SECONDARY OUTCOMES:
Phase 2: Overall Survival (OS) | 12 months after the first infusion of CD19-STAR-T cells
  OS is defined as the time from CD19-STAR-T cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.
Phase 2: Progression Free Survival (PFS) | 12 months after the first infusion of CD19-STAR-T cells
  PFS is defined as the time from the CD19-STAR-T cells infusion date to the date of disease progression assessed by investigators and based on the Lugano 2014 assessment criterion, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Phase 2: Time to response (TTR) | 12 months
  TTR is defined as the time from CD19-STAR-T infusion to first assessed CR or PR by investigators and based on the Lugano 2014 assessment criterion.
Phase 2: Duration of Response (DOR) | 12 months
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators and based on the Lugano 2014 assessment criterion for r/r B-cell NHL, or death regardless of cause.
Pharmacokinetics: Number and copy number of CD19-STAR-T cells (phase 1 and phase 2) | 12 months
  Number and copy number of CD19-STAR-T cells were assessed by number in peripheral blood. Blood samples were collected before and one year after cell infusion (until CD19-STAR-T cells were not detected for two consecutive times) to detect the number and copy number of CD19-STAR-T cells, and to evaluate the pharmacokinetics of CD19-STAR-T.
Pharmacokinetics: Persistence of CD19-STAR-T (phase 1 and phase 2) | 12 months
  Persistence of CD19-STAR-T cell assessed by number in peripheral blood.
Pharmacodynamics: Peak level of cytokines in serum (phase 1 and phase 2) | Up to 28 days after infusion
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), C reactive protein (CRP), ferritin. Peak was defined as the maximum post-baseline level of the cytokine.

OTHER OUTCOMES:
Relationship between infusion dose of CD19-STAR-T cells and efficacy | 12 months
  Peripheral blood was collected at the day of infusion (day 1), day 4, day 7, day 11, day 14, day 28, at least once every month after 28 days, at least once every three months after half a year, and at least once every six months after a year. The researchers will analyze the relationship between the number of CD19-STAR-T cells, copy number, cytokines level, and efficacy of CD19-STAR-T cells. The number of STAR-T cells was detected by flow cytometry, and the copy number was detected by quantitative PCR (qPCR).
To analyze the dynamic changes of STAR-T cells after infusion | 12 months
  The dynamic changes of the number and copy number of STAR-T cells in patients after CD19-STAR-T treatment were analyzed. To summarize the characteristic of the peak, expansion pattern, continuous expansion time and evolution of STAR-T cells in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Ph.D, Principal Investigator — Biotherapeutic Department, Chinese PLA General Hospital
Locations (2):
- China (2):
  - Biotherapeutic Department, Chinese PLA General Hospital, Beijing, Beijing Municipality
  - School of medicine, Tsinghua University & Changping Laboratory, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No